CLINICAL TRIAL: NCT04866303
Title: Protecting Our Community: A Pragmatic Randomized Trial of Home-Based COVID-19 Testing With Native American and Latino Communities
Brief Title: Protecting Our Community: COVID-19 Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); University of Washington (Other); Fred Hutchinson Cancer Center (Other); Salish Kootenai College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 5P20GM104417 (NIH); 5P20GM104417 (NIH)
Record Dates: First submitted 2021-04-27; First posted 2021-04-29 (Actual); Results first posted 2023-08-30 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: SARS-CoV-2; Covid19
Keywords: SARS-CoV-2; COVID-19; home-based testing; at home testing
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: A two-arm pragmatic randomized trial of SARS-CoV-2 home-based testing kit completion using active kit delivery by community health educators vs. passive kit delivery via mail.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active delivery (Experimental): For the participants randomized to the active arm will have their home collection kit registered on their behalf by bilingual (Spanish and English) community health workers, who are trusted community members. Home testing kits augmented with study developed materials will direct participants to contact the study team for assistance.
  Interventions: Diagnostic Test: Home-based SARS-CoV-2 test kit
- Passive delivery (Experimental): Participants randomized to the passive arm will receive a home test kit augmented with instructions on how to self-register their kit online, and will be directed to contact Everlywell for assistance, if needed.
  Interventions: Diagnostic Test: Home-based SARS-CoV-2 test kit

INTERVENTIONS:
Diagnostic Test: Home-based SARS-CoV-2 test kit — A two-arm pragmatic randomized trial of SARS-CoV-2 home-based testing kit completion using active kit assistance by community health educators vs. passive kit delivery. Will be done with two partner communities, Yakima Valley Latino community in WA and Flathead Reservation, American Indian community in MT. N = 200 participants in each community.

SUMMARY:
The COVID-19 pandemic has disproportionately affected American Indian (AI) and Latino communities, and these groups also have increased risk of poor prognosis due to high rates of chronic disease such as diabetes, cardiovascular disease, and cancer. In the northwestern United States, AI and Latino communities already face significant disparities in health care access, which have been further exacerbated by the COVID-19 pandemic. In the proposed study, Protecting Our Community: A Pragmatic Randomized Trial of Home-Based COVID Testing with Native American and Latino Communities, the investigators will leverage our long-term community-based participatory research partnerships to test the hypothesis that home-based testing will be feasible, impactful, and better-accepted using active delivery of test kits by trusted community health educators in two vulnerable, high-risk rural communities. Our two long-term partner communities are the Flathead Indian Reservation of the Confederated Salish and Kootenai Tribes in Montana, and the Yakima Valley of Washington, a large Latino community. The investigators will determine the cultural, social, behavioral, and economic barriers to home-based SARS-CoV-2 testing; culturally adapt and enhance home-testing educational materials and create home-testing instructional graphics and YouTube videos; conduct a 2-arm pragmatic randomized trial of active (delivered by community health educator) vs. passive (without community health educator) home-based testing kits (n = 200/community) for testing completion; and create a model for community-driven testing protocols that can have significant impact for increasing home-based testing uptake among AI and Latino communities nationally. This work will enable underserved AI and Latino communities to take full advantage of the coming wave of rapid point-of-care home tests and decrease the significant impact of COVID-19 in their communities.

DETAILED DESCRIPTION:
This clinical trial utilizes community-based participatory research partnerships to test the hypothesis that home-based testing for COVID-19 will be feasible, impactful, and better accepted using active assistance with the testing kits by trusted community members vs. passive delivery in two vulnerable high-risk rural communities. Our two long-term partner communities are the Flathead Indian Reservation of the Confederated Salish and Kootenai Tribes in Montana and the Yakima Valley of Washington, a large Hispanic community. The investigators will implement a two-arm pragmatic randomized trial during February to June 2021. Two hundred (200) adults per community will be randomized and stratified by age (18-25, 26-59, and 60+) to active vs. passive delivery. Our primary outcome will be the proportion of subjects who return testing collection kits in the active vs. passive arm. The trial will enable us to determine best practices and issues with home-based testing delivery in American Indian and Latino communities.

Participants randomized to both the active and passive arms will receive home testing kits augmented with materials developed by the study in both English and Spanish. In order to control for potential barriers to home testing kit delivery in this population (including internet access, digital literacy, English language proficiency) and limited access to mail delivery services (UPS, FedEx, etc.), participants in both study arms will be provided kit delivery and home collected sample return support coordinated by study staff. Coordination support options include (1) pick up / drop off at the research site, (2) shipping the home testing kit to the participant's mailing address by USPS or (3) home delivery/pick up to accommodate those with mobility concerns. The home testing kit selected in this study is the Everlywell COVID home-sampling kit.

Participants randomized to the passive arm will receive a home test kit with instructions on how to self-register their kit online, and will be directed to contact Everywell for assistance, if needed.

Participants randomized to the active arm will have their home collection kit registered on their behalf by community health workers while the participant remains on the phone. Study developed materials will direct participants to contact the study team for assistance.

Participants in both arms will receive study developed instructions to access their test results from the Everlywell online portal. Positive test results will be verbally provided by Everlywell contracted physicians. Study staff will confirm all participants have retrieved their test results from the online portal and referred to appropriate public health or clinical support as needed.

An initial survey of participant demographics and any current symptoms and medical conditions (including the RADx-UP Coordination and Data Collection Center common data & evaluation metrics) will be done via phone with participants prior to kit delivery.

Home testing kits returned and tested within 14 days of randomization will be considered "complete", while testing kits not returned or returned later than 14 days will be considered "not-complete". Within 14 days of randomization, will will conduct a phone delivered post-testing feedback survey with participants who completed their home testing kit to ask opinions on testing barriers and supports, interest in and barriers to self-testing before and after the study and usefulness of training materials. Participants who did not complete the home testing kit will be asked to provide reasons and barriers to completion. Post-testing feedback surveys will be brief and participants will receive a $35 gift card incentive for survey completion.

The investigators will also conduct in-depth, semi-structured, phone interview with 40 participants, 20 at each site, to collect perceptions of and experience with the home testing kit, vaccinations and other issues related to the pandemic. To facilitate collection of data at multiple timepoints in the study, interviews will be staggered. Interviews will occur roughly every two weeks over a 10-week period. The investigators will attempt to match interviews by active and passive arm assignment, completer and non-completer status, and timeframe. Twenty interviews with participants randomized to the active arm (10 participants who completed their home testing kits and 10 who did not) will be conducted as well as 20 interviews with participants randomized to the passive arm, also split evenly between participants who completed and not-completed their home testing kit. Participants who complete the in-depth, semi-structured phone interview will receive an incentive equal to $25.

Study consent, enrollment and study assessments will be conducted in the participant's preference of Spanish or English.

Harms

The investigators expect an extremely low occurrence of unfavorable events in this study and will be classifying negative study related harms to human subjects as either "social impacts", which for the purposes of this study are defined as an inadvertent and negative impact on an individual's standing in the community, within their family, their job, with the government, or with their finances as a result of participating in the study. Social impacts may also include worry (warranted or unwarranted), feeling upset or depressed, embarrassed, shameful, or guilty as a result of study participation or alternatively adverse events (AE) which are defined as any untoward medical occurrence in a subject during study participation.

Identification of both social impacts and AE will primarily be through passive surveillance, such as survey responses and conversations with site staff, and will be documented following informed consent until the final study assessment is complete. All social impacts and adverse events will be reported to the Data Safety Monitoring Board. Adverse events will be reported to the Montana State University IRB within 24 hours of site awareness. Study staff at each site will be trained in techniques to help resolve distress and connect participants to appropriate resources

Data Analysis and Sample Size Considerations

Our prior work with passive strategies has produced a return rate of approximately 70%.The investigators view a relative increase of 20% (absolute increase of 14%) to be a meaningful impact associated with the effort involved in active outreach, and therefore the investigators selected a sample with adequate power to detect such a difference. Specifically, with 400 total subjects (stratified by community) the study will have 90% power to detect an effect size associated with a rate ratio of 1.20, or an absolute difference of 14% (70% in passive, 84% in active). The investigators evaluated the design for robustness to assumptions regarding the passive return rate, and they have > 80% power to detect an absolute difference of 14% (relative rate of 1.23) if the passive return rate is 60%. No correction will be made for missing outcomes since the outcome is negative if no kit is returned. In addition, exploring the impact of using regression adjustment (logistic regression with an identity link) to account for community stratification, and the primary analysis maintains > 80% power for a range of passive rate differences across communities (ranging from 5% to 10%). All power calculations used the R statistical package and the PWR library and simulation methods.

The investigators will evaluate the net improvement in the rate of returning kits (primary outcome), comparing active vs. passive community outreach for uptake of home-based testing. Within each community, individuals will be randomized to active or passive delivery, and our primary analysis will compare the difference in the proportion of subjects who return collection kits while adjusting for community. Secondary analysis will compare active and passive rates across the communities to evaluate consistency of the intervention effect. Quantitative analysis of survey responses will focus on the creation of summary statistics that characterize the response to key survey items. An important statistical consideration is survey non-response and the potential for non-representative samples. The investigators will evaluate baseline factors that are potentially associated with non-response and then use inverse probability weighting (IPW) to correct for any potential bias associated with measured factors.

All statistical tests will be carried out at the 0.05 significance level, and estimates, 95% confidence intervals, and associated p-values will be reported for all tests. Analyses will be conducted using SAS 9.4 statistical software.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Member of study community
* No current significant symptoms consistent with COVID-19

Exclusion Criteria:

* < 18 years old
* Not a member of the study community
* Current significant symptoms consistent with COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra K Adams, MD, PhD, Principal Investigator — Montana State University
Locations (2):
- United States (2):
  - Salish Kootenai College, Pablo, Montana
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
In conjunction with tribal partners on the Flathead Reservation and at Salish Kootenai College in Montana, and with community partners in the Yakima Valley in Washington, we have developed a Data Sharing Plan. We will work closely with the Coordination and Data Collection Center (CDCC); the Social, Ethical, and Behavioral Implications program (SEBI); and the RADx-Up Consortium throughout the study to implement the Plan. All data will be deidentified and assigned an anonymous code by a member of the study team in each community before sharing with the broader study team for analysis. In addition, data collection instruments (including surveys, focus group and key informant interview questions, informed consent forms, community data collection tools, and educational material), deidentified coded data, and analyzed study trial results will be shared with the CDCC, SEBI, and RADx-UP Consortium.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While 273 participants were randomized, 268 were included in the analysis due to early withdraw or lost to follow-up
Period: Overall Study
Arm/Group | Passive Delivery | Active Delivery
Started (Total randomized) | 136 | 137
Withdrawal or Lost to Follow Up | 4 | 1
Completed | 132 | 136
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Population: Participants who provided consent and were randomized (both events happening on day 0). Baseline data not collected for 4 participants in the Passive Delivery Arm. Baseline data not collected for 1 participants in the Active Delivery Arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Passive Delivery | Active Delivery | Total
Number analyzed (Participants) | 136 | 137 | 273
Age, Customized [Count of Participants; unit: Participants] — Population: Baseline data not collected for 4 participants in the Passive Delivery Arm, Baseline data not collected for 1 participants in the Active Delivery Arm
  Participants
    18-25 years old: number analyzed (Participants) | 132 | 136 | 268
    18-25 years old | 17 | 16 | 33
    26-59 years old: number analyzed (Participants) | 132 | 136 | 268
    26-59 years old | 96 | 101 | 197
    60+ years old: number analyzed (Participants) | 132 | 136 | 268
    60+ years old | 19 | 19 | 38
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Baseline data not collected for 4 participants in the Passive Delivery Arm. Baseline data not collected for 1 participants in the Active Delivery Arm
  Participants
    Male: number analyzed (Participants) | 132 | 136 | 268
    Male | 22 | 27 | 49
    Female: number analyzed (Participants) | 132 | 136 | 268
    Female | 110 | 106 | 216
    Missing: number analyzed (Participants) | 132 | 136 | 268
    Missing | 0 | 3 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Baseline data not collected for 4 participants in the Passive Delivery Arm. Baseline data not collected for 1 participants in the Active Delivery Arm
  Participants
    Native American or Alaska Native: number analyzed (Participants) | 132 | 136 | 268
    Native American or Alaska Native | 28 | 32 | 60
    Hispanic or Latino: number analyzed (Participants) | 132 | 136 | 268
    Hispanic or Latino | 104 | 103 | 207
    Non-Hispanic White: number analyzed (Participants) | 132 | 136 | 268
    Non-Hispanic White | 9 | 9 | 18
Region of Enrollment [Number; unit: participants] — Population: Baseline data not collected for 4 participants in the Passive Delivery Arm. Baseline data not collected for 1 participants in the Active Delivery Arm
  participants
    United States: number analyzed (Participants) | 132 | 136 | 268
    United States | 132 | 136 | 268
Rural-Urban Commuting Area (RUCA) [Count of Participants; unit: Participants] — Population: Baseline data not collected for 4 participants in the Passive Delivery Arm. Baseline data not collected for 1 participants in the Active Delivery Arm
  Participants
    number analyzed (Participants) | 132 | 136 | 268
    Metropolitan | 17 | 10 | 27
    Micropolitan | 77 | 88 | 165
    Small town | 21 | 15 | 36
    Rural | 17 | 23 | 40
Education [Count of Participants; unit: Participants] — Population: Baseline data not collected for 4 participants in the Passive Delivery Arm. Baseline data not collected for 1 participants in the Active Delivery Arm
  Participants
    number analyzed (Participants) | 132 | 136 | 268
    No formal education | 2 | 2 | 4
    Elementary school | 14 | 14 | 28
    Some high school | 19 | 24 | 43
    High school degree or GED | 28 | 21 | 49
    Tech school | 4 | 5 | 9
    Some college | 28 | 26 | 54
    College degree | 13 | 19 | 32
    Graduate school degree | 2 | 3 | 5
    Missing | 22 | 22 | 44
Location [Count of Participants; unit: Participants] — Population: Baseline data not collected for 4 participants in the Passive Delivery Arm. Baseline data not collected for 1 participants in the Active Delivery Arm
  Participants
    number analyzed (Participants) | 132 | 136 | 268
    Flathead Reservation | 33 | 35 | 68
    Yakima Valley | 99 | 101 | 200

OUTCOME MEASURES:

1. Primary Outcome: SARS-CoV-2 Home-testing Kit Completion Active vs. Passive Arms
Description: Comparing the completed and successfully-completed test kits by study arm (randomization to either the active or passive arm)
Time Frame: 14 days from randomization for both completed and successfully-completed measurements
Population: 273 participants were both consented and randomized. 5 participants were lost to follow-up and excluded from analysis. An additional measure was added to make this more clear
Measure: Count of Participants; unit: Participants
Arm/Group | Passive Delivery | Active Delivery
Number analyzed (Participants) | 132 | 136
Participants
  Completed (kit arrived at processing lab) | 75 | 94
  Not-Completed (kit did not arrive at processing lab) | 57 | 42
Statistical Analysis 1: Comparison: Passive Delivery vs Active Delivery; Minimum testing kit completion rate of 70% in the passive study arm, and calculated that 400 total subjects would provide us with 90% power to detect an effect size associated with a rate ratio of 1.20, or an absolute difference of 14% (70% in passive, 84% in active). A futility boundary of 60% was identified by Community Advisory Board members as justification to prematurely halt trial enrollment if, after completing 25% of expected enrollment, successful test completion fell below that rate; Test type: Other — unadjusted logistic regression model; p = 0.04, Regression, Logistic; Odds Ratio (OR) = 1.79, 95% CI 2-sided [1.03 to 2.80]

2. Primary Outcome: SARS-CoV-2 Home-testing Kit Successfully-Completed Active vs. Passive Arms
Description: SARS-CoV-2 Home-testing Kit successfully-completed by study arm (randomization to either the active or passive arm)
Time Frame: 14 days from randomization for both completed and successfully-completed measurements
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Passive Delivery | Active Delivery
Number analyzed (Participants) | 132 | 136
Participants
  Successfully-Completed (kit was processed at lab, yielding a positive or negative result) | 61 | 74
  Unsuccessful-Completed (kit was not processed at lab due to sample effort) | 71 | 62
Statistical Analysis 1: Comparison: Passive Delivery vs Active Delivery; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.18, Regression, Logistic; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.86 to 2.26]

3. Post Hoc Outcome: SARS-CoV-2 Home-testing Kit Completion vs. Successful Rates Across the Communities
Description: SARS-CoV-2 Home-testing Kit Completed vs. Successful completed rates, stratified by community.
Time Frame: 14 days from randomization for both completed and successfully-completed measurements
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Passive Delivery | Active Delivery
Number analyzed (Participants) | 132 | 136
Participants
  Yakima Valley, Not-Completed | 39 | 31
  Yakima Valley, Completed-Not Successful | 13 | 14
  Yakima Valley, Completed-Successful | 47 | 56
  Flathead, Not-Completed | 18 | 11
  Flathead, Completed-Not Successful | 1 | 6
  Flathead, Completed-Successful | 14 | 18

ADVERSE EVENTS:
Time Frame: Adverse experiences (adverse events and social impacts) were collected from day 0 through the last study assessment or day 21, whichever occurred first.
Description: In addition to the clinicaltrials.gov definition of adverse event, we also included a breakdown of safety procedures in our adverse event definition. Social impacts were defined as (1) inadvertent and negative impact on an individual's standing in the community, within their family, their job, with the government, or with their finances as a result of participating in the study. Adverse experiences were identified through surveys, and per protocol conversations & study assessments.
Arm/Group | Passive Delivery | Active Delivery
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/137
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/137
Other Adverse Events (participants affected / at risk) | 0/132 | 1/136
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Passive Delivery (N=132) | Active Delivery (N=136)
Social Impacts (Social circumstances) | 0 (0) | 1 (1) — Inadvertent and negative impact on an individual's standing in the community, within their family, their job, with the government, or with their finances as a result of participating in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Flathead Tribal Council expects prior approval for any secondary usage of Tribal data uploaded to RADx-UP central repository and coordinating center and maintains the authority to review all publications, conference presentations and other scholarly works prior to dissemination.

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT04866303/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT04866303/SAP_001.pdf